CLINICAL TRIAL: NCT00993460
Title: Diacylglycerols and Insulin Action in Skeletal Muscle Upon Caloric Restriction
Brief Title: Study of Changes in Skeletal Muscle After Caloric Restriction
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Charles R. Flynn, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: IRB #091145
Record Dates: First submitted 2009-10-07; First posted 2009-10-12 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Obesity; Insulin sensitivity; Inflammation
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, muscle tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal body weight: Female subjects, ages 21-65 yrs, with BMI of 21-27 kg/m2 with normal glucose tolerance.
- Roux-en-Y gastric bypass: Female subjects ages 21-65 with insulin resistance and scheduled for Roux-en-Y gastric bypass at Vanderbilt University Medical Center will be studied before and 4-6 weeks after surgery.

SUMMARY:
Research has shown that fat stored within muscles affects the muscle's sensitivity to insulin and ability to handle blood glucose. The purpose of this study is to examine the effects of weight loss surgery-induced caloric restriction on the accumulation and types of fats within skeletal muscle, as well as the effects of such caloric restriction on insulin sensitivity and inflammatory responses in skeletal muscle. The investigator proposes that caloric restriction will result in decreases in diacylglycerols enriched with saturated fat and increases in diacylglycerols enriched with monounsaturated fats.

DETAILED DESCRIPTION:
We hypothesize that in a setting of surgically-induced weight loss decrements in select DAGs result in improved glucose utilization, altered insulin signaling and decreased inflammatory responses. We propose to examine the impact of molecular DAG species accumulation on glucose utilization, insulin signaling and inflammation in skeletal muscle from morbidly obese subjects before/after 10% weight loss facilitated by Roux-en-Y Gastric Bypass (RYGB). We will compare these results to those from a control, normal weight cohort

The detected differences in DAG molecular species, insulin action, inflammatory responses between normal and obese subjects (before/after weight loss) will emphasize pathways coordinately altered as a consequence of adiposity and RYGB surgery. The primary endpoints for this study will be: Insulin sensitivity (glucose Rd, insulin levels, DAG mass, DAG species amounts).Secondary endpoints will be: FFA levels, inflammatory cytokine production, and insulin signaling in skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* For Normal Weight Subjects:

  * Age 21-65 years
  * BMI of 21 to 27 kg/m2
  * Normal glucose tolerance as determined by OGTT on day of screening
  * No family history of diabetes
* For Morbidly Obese Subjects:

  * Age 21-65 years
  * BMI of 30 to 65 kg/m2
  * Scheduled for Roux-en-Y gastric bypass at Vanderbilt Medical Center
  * Insulin resistant as determined by OGTT on day of screening

Exclusion Criteria (for all subjects):

* Clinically significant heart disease
* Clinically significant hepatic or renal disease
* Pregnancy
* Breastfeeding
* Any abnormality that would preclude safe completion of study
* Use of statins
* Use of thiazide or furosemide diuretics, beta blockers, or other chronic medications with known adverse effects on glucose tolerance levels unless subject has been on stable dose of such medications for the past 3 months before entering the study

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female subjects approved for Roux-en-Y gastric bypass surgery at Vanderbilt University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
UPLC-ESI MS/MS profiling of lipd extracts from muscle biopsies to evaluate effects of gastric bypass induced-caloric restriction on diacylglycerol molecular species accumulation. | 1 year

SECONDARY OUTCOMES:
To evaluate the effects of gastric bypass induced-caloric restriction on skeletal muscle insulin action via a hyperinsulinemic-euglycemic clamp and profiling markers of insulin signaling. | 1 year
To evaluate the effects of gastric bypass induced-caloric restriction on lipid-mediated inflammatory responses by profiling cytokines and free fatty acids in blood and inflammation markers in skeletal muscle biopsies. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Flynn, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji Abumrad, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States